CLINICAL TRIAL: NCT02665416
Title: An Open-Label, Multicenter, Dose Escalation Phase Ib Study With Expansion Cohorts to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics, and Therapeutic Activity of RO7009789 (CD40 Agonistic Monoclonal Antibody) in Combination With Vanucizumab (Anti-Ang2 and Anti-VEGF Bi-Specific Monoclonal Antibody, Part I) or Bevacizumab (Anti-VEGF Monoclonal Antibody, Part II) in Patients With Metastatic Solid Tumors
Brief Title: Study Evaluating the Safety, Pharmacokinetics (PK), Pharmacodynamics (PD), and Therapeutic Activity of Selicrelumab (RO7009789) With Vanucizumab or Bevacizumab in Participants With Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BP29889; 2015-003480-11 (EudraCT Number); RG7876 (Other: Roche)
Record Dates: First submitted 2016-01-15; First posted 2016-01-27 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Advanced/Metastatic Solid Tumors
MeSH Terms: interventions — selicrelumab; vanucizumab; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part I: Selicrelumab, Vanucizumab/Bevacizumab (Experimental): Participants will receive a fixed dose of vanucizumab, 2 grams via IV infusion on Days 1 and 15 of every 28-day cycle. Selicrelumab will be given SC in ascending dose levels on Day 2 of Cycles 1 to 4 and every third cycle thereafter. Treatment will continue as long as the participant experiences clinical benefit or until unacceptable toxicity, withdrawal of consent, or the end of Part I of the study (expected 24 months). Due to the discontinuation of Vanucizumab development, Participants ongoing in Part I will switch from Vanucizumab to Bevacizumab. All the dose escalation has been performed using Vanucizumab.
  Interventions: Drug: Selicrelumab; Drug: Vanucizumab
- Part II: Selicrelumab, Bevacizumab (Experimental): Bevacizumab will be administered via IV infusion on days 1 and 15 of every 28-day cycle. Selicrelumab will be given SC after the Bevacizumab infusion at the dose determined in the Part I of the study on Day 2 of Cycles 1 to 4 and every third cycle thereafter. Treatment will continue as long as the participant experiences clinical benefit or until unacceptable toxicity, withdrawal of consent, or the end of Part II of the study (expected 18 months).
  Interventions: Drug: Selicrelumab; Drug: Bevacizumab

INTERVENTIONS:
Drug: Selicrelumab — Selicrelumab will be provided as concentrate for solution to be administered via SC injection
  Other Names: RO7009789
Drug: Vanucizumab — Vanucizumab will be provided as solution to be administered via IV infusion.
  Arms: Part I: Selicrelumab, Vanucizumab/Bevacizumab
Drug: Bevacizumab — Bevacizumab will be administered via IV infusion.
  Arms: Part II: Selicrelumab, Bevacizumab

SUMMARY:
This open-label, two-part study is designed to assess the safety, PK, PD, and therapeutic activity of Selicrelumab in combination with vanucizumab or bevacizumab in participants with metastatic solid tumors not amenable to standard treatment. Part I (dose escalation) is designed to establish the maximum tolerated dose (MTD) of Selicrelumab in this combination. Part II (expansion) is intended to characterize the safety and tolerability of Selicrelumab in combination with bevacizumab among indication-specific cohorts and to confirm the recommended dose.

ELIGIBILITY:
Inclusion Criteria:

* Part I: Histologically confirmed advanced/metastatic solid tumor (except prostate cancer and squamous non-small cell lung cancer [NSCLC])
* Part II: Histologically confirmed advanced/metastatic platinum-resistant ovarian carcinoma (aPROC), head and neck squamous cell carcinoma (HNSCC), or non-squamous NSCLC previously treated with anti-PD-L1/PD-1 inhibitor alone or in combination (e.g. atezolizumab, nivolumab, pembrolizumab, durvalumab, avelumab)
* Checkpoint inhibitor (CPI)- experienced patients must have experienced documented disease progression on or after PD-L1/PD-1 inhibitor therapy
* In CPI-experienced patients, the PD-L1/PD-1 inhibitor must have been part of the most recent systemic anticancer therapy administered prior to study enrollment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Life expectancy >/= 16 weeks
* Adequate hematologic, renal, hepatic, and cardiovascular function
* Measurable disease per Response Evaluation Criteria in Solid Tumors, v 1.1 (RECIST v1.1)
* Tumors must be acceptable for biopsy. Participants in Part II may be enrolled without a biopsy if the collection is not clinically feasible.
* Agreement to use adequate contraceptive measures among men or among women of childbearing potential

Exclusion Criteria:

* Prostate cancer or squamous NSCLC
* Recent systemic anti-cancer treatment
* Prior treatment with anti-programmed death (PD) 1 or anti-programmed death ligand (PD-L) 1 therapeutic antibody, vanucizumab, or compounds targeting cluster of differentiation (CD) 40 less than 4 weeks or 5xt1/2 (whichever is shorter) prior to enrollment
* Part II: Treatment targeting vascular endothelial growth factor (VEGF) or receptor within 12 months prior to enrollment
* Systemic immunosuppressive medication within 2 weeks prior to day 1 of cycle 1
* Chronic daily treatment with non-steroidal anti-inflammatory drugs
* Unacceptable/unresolved toxicity from prior anti-cancer therapy
* Patients who have had a surgical procedure or significant traumatic injury within 28 days prior to initiation of study treatment, or a core biopsy or other minor surgical procedure within 7 days prior to initiation of study treatment
* Bisphosphonate therapy for symptomatic hypercalcemia
* Significant vascular disease
* History of hypertensive crisis or hypertensive encephalopathy
* Current or recent use of aspirin (>325 mg/day) or clopidogrel (>75 mg/day)
* History of vein thrombosis/thromboembolism, or use of anticoagulants within 7 days prior to study drug
* Primary tumor in place in participants with colorectal cancer, or evidence of bowel involvement (metastasis, direct tumor invasion) in participants with other non-gastrointestinal cancer
* Significant cardiovascular or cerebrovascular disease within 6 months prior to D1 of C1
* History of fistula, bowel obstruction, perforation, or abscess
* Prior radiotherapy to pelvis or abdomen, recto-sigmoid involvement, or bowel involvement among participants with aPROC
* Severe non-healing wound, active ulcer or untreated bone fracture
* Pregnant or lactating women
* History of autoimmune disease
* Human immunodeficiency virus (HIV) or hepatitis B or C
* Severe infection or receipt of a live/attenuated vaccine within 4 weeks prior to D1 of C1
* Other significant malignancies within 3 years prior to D1 of C1
* Allergy/hypersensitivity to study drug
* Prior allogeneic bone marrow or solid organ transplant
* Other conditions/findings that may contraindicate use of study drug
* Major surgery within 4 weeks prior to study drug
* Known clinically significant liver disease
* History of hemoptysis or bleeding diathesis, or known coagulopathies
* Known symptomatic or untreated central nervous system (CNS) malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Dose-Limiting Toxicities (DLTs) | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  From Day (D) 1 until D28 of Cycle (C)1 (cycle length=28 days)
MTD of Selicrelumab in Combination With Vanucizumab | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  From D1 until D28 of C1 (cycle length=28 days)
Recommended Phase II Dose of Selicrelumab in Combination With Vanucizumab | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  From D1 until D28 of C1 (cycle length=28 days)
Percentage of Participants With Adverse Events (AEs) | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  From D1 of C1 until treatment discontinuation and approximately 45 days after last dose (cycle length=28 days)
Part II: Clinical Activity of SC Selicrelumab in Combination with Bevacizumab as Assessed by Response Evaluation in Solid Tumors, Version 1.1 (RECIST v1.1) | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  From D1 of C1 through safety follow up visit (45 days post final dose; Cycle = 28 days)
Part II: Percentage of Participants With Best Overall Response per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) Criteria | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Tumor assessments at Screening and on D1 of C3, C5, C7; and every 12 weeks thereafter until disease progression (cycle length=28 days)
Part II: Duration of Objective Response per RECIST v1.1 Criteria | TBaseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Tumor assessments at Screening and on D1 of C3, C5, C7; and every 12 weeks thereafter until disease progression (cycle length=28 days)
Part II: Percentage of Participants With Disease Control per RECIST v1.1 Criteria | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Tumor assessments at Screening and on D1 of C3, C5, C7; and every 12 weeks thereafter until disease progression (cycle length=28 days)
Part II: Progression-free Survival (PFS) per RECIST v1.1 Criteria | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Tumor assessments at Screening and on D1 of C3, C5, C7; and every 12 weeks thereafter until disease progression (cycle length=28 days)

SECONDARY OUTCOMES:
Percentage of Participants With Anti-Drug Antibodies (ADAs) to Selicrelumab | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Predose (-1 hour [h]) on D2 of C1, C2, C3, C4, C7, and every 3 cycles until/at disease progression and/or 45 days after last dose (cycle length=28 days)
Percentage of Participants with ADAs to Vanucizumab | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Predose (within 10 minutes [min] before infusion) on D1 of C1, C2, C4, and every 2 cycles until/at disease progression and/or 45 days after last dose (cycle length=28 days)
Area Under the Concentration-Time Curve From Time 0 to Last Measureable Concentration (AUClast) of Selicrelumab Following Subcutaneous (SC) Administration | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Predose (-1 h) and 3 (only C2), 4, 8, 24, 48, 72 h postdose on C1 and C2; predose (-1 h) and 8 h postdose on C3, C4, C7, and every 3 cycles until/at disease progression and/or 45 days after last dose (up to 24 months in Part I and 18 months in Part II; cycle length=28 days)
Area Under the Concentration-Time Curve From Time 0 to Infinity (AUCinf) of Selicrelumab Following SC Administration | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Predose (-1 h) and 3 (only C2), 4, 8, 24, 48, 72 h postdose on C1 and C2; predose (-1 h) and 8 h postdose on C3, C4, C7, and every 3 cycles until/at disease progression and/or 45 days after last dose (cycle length=28 days)
Maximum Concentration (Cmax) of Selicrelumab Following SC Administration | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Predose (-1 h) and 3 (only C2), 4, 8, 24, 48, 72 h postdose on C1 and C2; predose (-1 h) and 8 h postdose on C3, C4, C7, and every 3 cycles until/at disease progression and/or 45 days after last dose (cycle length=28 days)
Time to Maximum Concentration (Tmax) of Selicrelumab Following SC Administration | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Predose (-1 h) and 3 (only C2), 4, 8, 24, 48, 72 h postdose on C1 and C2; predose (-1 h) and 8 h postdose on C3, C4, C7, and every 3 cycles until/at disease progression and/or 45 days after last dose (cycle length=28 days)
Apparent Clearance (CL/F) of Selicrelumab Following SC Administration | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Predose (-1 h) and 3 (only C2), 4, 8, 24, 48, 72 h postdose on C1 and C2; predose (-1 h) and 8 h postdose on C3, C4, C7, and every 3 cycles until/at disease progression and/or 45 days after last dose (cycle length=28 days)
Apparent Volume of Distribution (Vd/F) of Selicrelumab Following SC Administration | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Predose (-1 h) and 3 (only C2), 4, 8, 24, 48, 72 h postdose on C1 and C2; predose (-1 h) and 8 h postdose on C3, C4, C7, and every 3 cycles until/at disease progression and/or 45 days after last dose (cycle length=28 days)
Apparent Terminal Half-Life (t1/2) of Selicrelumab Following SC Administration | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Predose (-1 h) and 3 (only C2), 4, 8, 24, 48, 72 h postdose on C1 and C2; predose (-1 h) and 8 h postdose on C3, C4, C7, and every 3 cycles until/at disease progression and/or 45 days after last dose (cycle length=28 days)
Part I: AUClast of Vanucizumab | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Predose (within 10 min) on D1 of C1, C2, C4, C6, C8, every 2 cycles thereafter disease progression and/or 45 days after last dose; predose (within 10 min), end of infusion (infusion duration=60-90 min) on D15 of C1 to C9 and each cycle thereafter until disease progression and/or 45 days after last dose; 6 and 24 h postdose on D15 of C1 and C8 (cycle length = 28 days)
Part I: AUCinf of Vanucizumab | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Predose (within 10 min) on D1 of C1, C2, C4, C6, C8, every 2 cycles thereafter disease progression and/or 45 days after last dose; predose (within 10 min), end of infusion (infusion duration=60-90 min) on D15 of C1 to C9 and each cycle thereafter until disease progression and/or 45 days after last dose; 6 and 24 h postdose on D15 of C1 and C8 (cycle length = 28 days)
Part I: Concentration at the End of Infusion (Cend) of Vanucizumab | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Predose (within 10 min) on D1 of C1, C2, C4, C6, C8, every 2 cycles thereafter disease progression and/or 45 days after last dose; predose (within 10 min), end of infusion (infusion duration=60-90 min) on D15 of C1 to C9 and each cycle thereafter until disease progression and/or 45 days after last dose; 6 and 24 h postdose on D15 of C1 and C8 (cycle length = 28 days)
Part I: CL of Vanucizumab | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Predose (within 10 min) on D1 of C1, C2, C4, C6, C8, every 2 cycles thereafter disease progression and/or 45 days after last dose; predose (within 10 min), end of infusion (infusion duration=60-90 min) on D15 of C1 to C9 and each cycle thereafter until disease progression and/or 45 days after last dose; 6 and 24 h postdose on D15 of C1 and C8 (cycle length = 28 days)
Part I: Vss of Vanucizumab | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Predose (within 10 min) on D1 of C1, C2, C4, C6, C8, every 2 cycles thereafter disease progression and/or 45 days after last dose; predose (within 10 min), end of infusion (infusion duration=60-90 min) on D15 of C1 to C9 and each cycle thereafter until disease progression and/or 45 days after last dose; 6 and 24 h postdose on D15 of C1 and C8 (cycle length = 28 days)
Part I: t1/2 of Vanucizumab | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Predose (within 10 min) on D1 of C1, C2, C4, C6, C8, every 2 cycles thereafter disease progression and/or 45 days after last dose; predose (within 10 min), end of infusion (infusion duration=60-90 min) on D15 of C1 to C9 and each cycle thereafter until disease progression and/or 45 days after last dose; 6 and 24 h postdose on D15 of C1 and C8 (cycle length = 28 days)
Part I: Percentage of Participants With Best Overall Response per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) Criteria | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Tumor assessments at Screening and on D1 of C3, C5, C7; and every 12 weeks thereafter until disease progression (cycle length=28 days)
Part I: Duration of Objective Response per RECIST v1.1 Criteria | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Tumor assessments at Screening and on D1 of C3, C5, C7; and every 12 weeks thereafter until disease progression (cycle length=28 days)
Part I: Percentage of Participants With Disease Control per RECIST v1.1 Criteria | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Tumor assessments at Screening and on D1 of C3, C5, C7; and every 12 weeks thereafter until disease progression (cycle length=28 days)
Part I: Progression-free Survival (PFS) per RECIST v1.1 Criteria | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Tumor assessments at Screening and on D1 of C3, C5, C7; and every 12 weeks thereafter until disease progression (cycle length=28 days)
Part I: Clinical Activity of SC Selicrelumab in Combination with Bevacizumab as Assessed by Response Evaluation in Solid Tumors, Version 1.1 (RECIST v1.1) | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  From D1 of C1 through safety follow up visit (45 days post final dose; cycle length = 28 days)
Change in Blood and Tumor Tissue Immune Cell Subpopulations | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Part I: C1 at D1 pre-dose Vanicizumab, D4, D9 (D15 pre and 6h post for cohorts 8 onwards); C2 at D1 and D9; C4,7,10 at D1 and D9; PD Part II: C1 D1(pre), D3,D8,D15; C2,4,7,10 D1,D8; PD
Change in Peripheral Blood Level of Cytokines | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  C1D1 pre-dose Vanicizumab, C1 D2 pre-dose Selicrelumab and 3h post-dose Selicrelumab, C2D1 pre-dose Vanicizumab, C2D2 pre-dose Selicrelumab and 3h post-dose Selicrelumab, C4 D2 pre-dose Selicrelumab and 3h post-dose, PD
Change in Blood Soluble Proteins | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  D1, 2, 3, 9, 15 of C1; D1, 3, 9, 15 of C2; D1 of C 4,5; D1, 15 of C7, D1 of C10, PD
Percentage of Participants With Best overall Response Immune-Related Response Criteria (irRC) | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Tumor assessments at Screening and on D1 of C3, C5, C7; and every 12 weeks thereafter until disease progression (cycle length=28 days)
Duration of Objective Response per irRC | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Tumor assessments at Screening and on D1 of C3, C5, C7; and every 12 weeks thereafter until disease progression (cycle length=28 days)
Percentage of Participants With Disease Control per irRC | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Tumor assessments at Screening and on D1 of C3, C5, C7; and every 12 weeks thereafter until disease progression (cycle length=28 days)
PFS per irRC | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  Tumor assessments at Screening and on D1 of C3, C5, C7; and every 12 weeks thereafter until disease progression (cycle length=28 days)
Clinical Activity of SC Selicrelumab in Combination with Bevacizumab as Assessed by Unidimensional Immune-Related Response Criteria (irRC) | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  From D1 of C1 through safety follow up visit (45 days post final dose; cycle length = 28 days)
Overall Survival (OS) | Baseline until Participant's discontinuation or death, whichever occurs first (up to approximately 42 months)
Concentration at the end of Infusion (Cend) of Bevacizumab | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  D1 and D15 of C1, then D1 of every cycle until C7; at radiographical disease progression/tumor regression; at safety follow up visit (45 days post final dose; Cycle = 28 days)
Minimum Concentration (Cmin) of Bevacizumab after Infusion | Baseline until Participant's discontinuation or death, whichever occurs first, as per schedule in the description (up to approximately 42 months)
  D1 and D15 of C1, then D1 of every cycle until C7; at radiographical disease progression/tumor regression; at safety follow up visit (45 days post final dose; Cycle = 28 days)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (16):
- United States (5):
  - Cedars Sinai Medical Center, Los Angeles, California
  - Univ of CO Health Science Ctr, Denver, Colorado
  - Yale Cancer Center; Medical Oncology, New Haven, Connecticut
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
- Cliniques Universitaires St-Luc, Brussels, Belgium
- University Health Network; Princess Margaret Hospital; Medical Oncology Dept, Toronto, Ontario, Canada
- Rigshospitalet; Onkologisk Klinik, København Ø, Denmark
- Irccs Ospedale San Raffaele;Oncologia Medica, Milan, Lombardy, Italy
- Netherlands (2):
  - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - Erasmus Medisch Centrum, Rotterdam
- Spain (5):
  - ICO L'Hospitalet; Servicio de oncologia medica, L'Hospitalet de Llobregat, Barcelona
  - Hospital del Mar; Servicio de Oncologia, Barcelona
  - Hospital Univ Vall d'Hebron; Servicio de Oncologia, Barcelona
  - START Madrid. Centro Integral Oncologico Clara Campal; CIOCC, Madrid
  - Hospital Clinico Universitario de Valencia; Servicio de Onco-hematologia, Valencia